CLINICAL TRIAL: NCT00234234
Title: Predictors of the Response to Adalimumab in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/145/HP
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Biologics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory rheumatic disease which is characterized by joint inflammation (clinical involvement), by osteo-cartilaginous lesions (structural damage) and generally by bone involvement. All those features lead to great disability. Because it represents a major problem of the public health care system, RA has been selected as one of the main objectives of the government for the next five years.

RA patients who do not respond to DMARDs require a treatment by TNF-a blocking agents. However, no information is available to predict the clinical, structural and bone responses to those new drugs that can be responsible of severe side-effects. Moreover, they are particularly expensive since their yearly cost is estimated between 75000 and 112500 k euros for the G4 region.

The purpose of the present research project is to determine potential predictive factors of the response to a new TNF-a blocker ie adalimumab. To address this question, several investigations will be performed including measurement of different blood markers, particularly bone markers, well-defined autoantibodies and new autoantibody populations identified by proteomic analysis, large-scale analysis of gene expression with cDNA arrays from blood mononuclear cells, and use of different imaging tools.

The criteria of judgement will be the clinical, structural and bone responses to those new agents.

This study requires the recruitment of about 100 patients receiving adalimumab for a 1-year period.

At the end of the study, we hope to identify predictive factors of the response to adalimumab, which will lead to a better management of this TNF-a blocker. Indeed, they will be prescribed only for the patients who are likely to respond to those drugs. Thus, this study should allow to elaborate theranostic algorithms. Such an approach will have great benefits for the patients: more rapid efficacy, less severe side-reactions and lower costs.

ELIGIBILITY:
Inclusion Criteria:

* ACR classification criteria of RA
* DAS 28 > 5.1
* inadequately controlled by at least one DMARD
* biologics naïve

Exclusion Criteria:

* exclusion criteria of adalimumab and methotrexate (regulation authorities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical response
Structural response : X-rays
Bone response : osteodensitometry

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Le Loët, MD, Pr Rheumatology, Principal Investigator — University Hospital, Rouen; Marcelli Christian, Study Director — University Hospital, Caen
Locations (1):
- MARCELLI, Caen, Basse Normandie, France

REFERENCES:
- [Derived] Vittecoq O, Guillou C, Hardouin J, Gerard B, Berenbaum F, Constantin A, Rincheval N, Combe B, Lequerre T, Cosette P. Validation in the ESPOIR cohort of vitamin K-dependent protein S (PROS) as a potential biomarker capable of predicting response to the methotrexate/etanercept combination. Arthritis Res Ther. 2022 Mar 21;24(1):72. doi: 10.1186/s13075-022-02762-5. PMID 35313956
- [Derived] Golinski ML, Vandhuick T, Derambure C, Freret M, Lecuyer M, Guillou C, Hiron M, Boyer O, Le Loet X, Vittecoq O, Lequerre T. Dysregulation of RasGRP1 in rheumatoid arthritis and modulation of RasGRP3 as a biomarker of TNFalpha inhibitors. Arthritis Res Ther. 2015 Dec 26;17:382. doi: 10.1186/s13075-015-0894-9. PMID 26714738
- [Derived] Ternant D, Ducourau E, Fuzibet P, Vignault C, Watier H, Lequerre T, Le Loet X, Vittecoq O, Goupille P, Mulleman D, Paintaud G. Pharmacokinetics and concentration-effect relationship of adalimumab in rheumatoid arthritis. Br J Clin Pharmacol. 2015 Feb;79(2):286-97. doi: 10.1111/bcp.12509. PMID 25223394
- [Derived] Blache C, Lequerre T, Roucheux A, Beutheu S, Dedreux I, Jacquot S, Le Loet X, Boyer O, Vittecoq O. Number and phenotype of rheumatoid arthritis patients' CD4+CD25hi regulatory T cells are not affected by adalimumab or etanercept. Rheumatology (Oxford). 2011 Oct;50(10):1814-22. doi: 10.1093/rheumatology/ker183. Epub 2011 Jul 26. PMID 21791546